CLINICAL TRIAL: NCT05612789
Title: Intervening on Frailty to Improve Outcomes for Older Allogeneic Transplant Recipients
Brief Title: Improve Outcomes for Older Allogeneic Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 07422; Penn IRB# 851615 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2022-10-21; First posted 2022-11-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Allogeneic Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Prehab) (Experimental): Pre-frail and frail subjects will attend at least twice weekly exercise sessions with a physical therapist and be given an exercise program to complete at home prior to admission for HCT. Patients enrolled in this cohort can continue on to Cohort B.
  Interventions: Behavioral: Exercise Program (Cohort A Prehab)
- Cohort B (Rehab) (Experimental): All patients 60 years and older upon discharge from their initial hospital stay for HCT will attend at least weekly exercise sessions with a physical therapist and be given an exercise program to complete at home with sessions continued through Day +100 after HCT.
  Interventions: Behavioral: Exercise Program (Cohort B Rehab)

INTERVENTIONS:
Behavioral: Exercise Program (Cohort A Prehab) — Pre-frail and frail potential HCT recipients 60 years and older will participate in a supervised exercise program from the time of enrollment up until HCT admission. Exercise compliance will be measured in part through physical activity trackers.from time of discharge from HCT until day +100 post-HCT. All HCT recipients 60 years and older will participate in a supervised exercise program from the time of discharge from HCT admission until day +100 post-HCT. Exercise compliance will be measured in part through physical activity trackers.
  Arms: Cohort A (Prehab)
Behavioral: Exercise Program (Cohort B Rehab) — All HCT recipients 60 years and older will participate in a supervised exercise program from the time of discharge from HCT admission until day +100 post-HCT. Exercise compliance will be measured in part through physical activity trackers.
  Arms: Cohort B (Rehab)

SUMMARY:
This is an interventional pilot study to determine whether implementation of a supervised exercise program can improve outcomes in subjects undergoing allogeneic HCT. The primary objective is to determine feasibility. Up to 60-72 evaluable subjects will be enrolled. Evaluable subjects are defined as those participating in the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

Cohort A (Prehab)

1. Age 60 years or older.
2. Planned allogeneic HCT in the next 1-6 months.
3. Hematological malignancy as the indication for HCT.
4. Pre-frail or frail by Fried frailty phenotype.

Cohort B (Rehab)

1. Age 60 years or older.
2. Planned allogeneic HCT or HCT within the last 30 days.
3. Hematological malignancy as the indication for HCT.

Exclusion Criteria:

Cohorts A and B

1. Comorbid disability or illness that prevents safe exercise.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled subjects who participate in the supervised exercise program | From 3 months prior to HCT to 100 days after HCT
Median number of exercise sessions delivered pre-HCT and post-HCT. | From 3 months prior to HCT to 100 days after HCT

SECONDARY OUTCOMES:
Hospital LOS for HCT | From date of randomization until the date of first documented discharge from the hospital, assessed up to 100 months
Rate of readmission | From time of discharge from initial hospital stay up through 1-2 years after HCT
6-month and 1-year overall mortality | From day 0 of HCT to 6 months and 1-year] 6. 1-year and 2-year OS
1-year and 2-year OS | From day 0 of HCT to 1-year and 2-years
1-year and 2-year PFS | From day 0 of HCT to 1-year and 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Shannon McCurdy, MD, Principal Investigator — Penn Medicine
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes